CLINICAL TRIAL: NCT01964794
Title: Improving Anticoagulant Therapy Through Warfarin Metabolite Profiling
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Collaborators: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 135288
Record Dates: First submitted 2013-10-09; First posted 2013-10-17 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Stable Target INR
Keywords: Warfarin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood specimens to identify coumadin genetic and metabolic biomarkers.

SUMMARY:
Clinically relevant biomarkers for warfarin identified in this study will provide crucial leads for subsequent studies to assess their predictive value during anticoagulant therapy. This knowledge will aid stratifying risk among patients to improve therapeutic outcomes and decrease adverse drug events and associated health care costs. Collectively, these efforts will provide a critical foundation for future research using a metabolite biomarker strategy in a clinical setting to revolutionize warfarin therapy. Through its application, a real-time assessment of warfarin metabolism for each patient could lead to a truly personalized dosing strategy and improve patient safety for this life-saving drug.

DETAILED DESCRIPTION:
Coumadin (R/S-warfarin) is a commonly prescribed anticoagulant for over 20 million Americans for the treatment of atrial fibrillation, mechanical heart valves, venous thromboembolism and other coagulopathies. While highly efficacious, warfarin treatment is challenging due to a narrow therapeutic range and high inter-individual variations in response. Optimal warfarin dosage relies on a potentially lengthy trial-and-error process to optimize dosage for a desired anticoagulant response as measured by the international normalization ratio (INR), a prothrombin test. Even when a maintenance dose is achieved, patients are prone to testing out of the target INR range, and thus are at risk of hemorrhaging (over-dosing) or thromboembolism (under-dosing). In fact, warfarin is among the top ten drug-related causes of serious adverse drug events and increased health care costs. The progressive increase in warfarin use necessitates a better understanding of the mechanisms underlying inter-individual variability in responses to anticoagulant therapy. Our long-term goal is to identify metabolic biomarkers correlating with clinical responses to warfarin therapy and then utilize this knowledge to predict safe and effective dosing for patients based on a single blood draw.

Therapeutic outcomes for patients involve a balance between warfarin dosing and its metabolism to maintain a stable target INR. There is an initial lengthy titration stage in which dosing is increased to achieve but not surpass a target INR range. The potency of this effect depends on warfarin metabolism, which counters the dosing effect on patients by inactivating the drug. Warfarin undergoes extensive metabolism through distinct enantio- and regio-specific metabolic pathways to yield a complex array of essentially inactive isomeric metabolites. Warfarin is clinically available as an equal mixture of R and S enantiomers. S-Warfarin is about four times more potent than R-warfarin, and presumably dominates the anticoagulant response to therapy. During maintenance dosing, a longer metabolic half-life for R-warfarin leads to higher accumulation levels in plasma than those observed for S-warfarin. Variations in R-and S-warfarin plasma levels may potentiate the anticoagulant effect of both drug isomers and the corresponding responses to therapy. For our exploratory study, we will identify biomarkers within patient metabolic profiles for R-and S-warfarin that predict clinical outcomes for the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 60 - 69 originally. Opened inclusion criteria age to include 18-79 years of age.
2. Potential participant received a warfarin maintenance dose with a stable INR (defined as within target range over a two month (60 day) period that includes a minimum of two clinical visits).
3. Potential participant has taken warfarin as prescribed over the past three days.

Exclusion Criteria:

1. Female
2. Potential participant receiving a warfarin while not achieving a stable INR (defined as within target range over a two month (60 day) period that includes a minimum of two clinical visits).
3. Potential participant has not received any warfarin over the past three days.

Ages: 60 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Originally, for this pilot study, we chose a sample population size of 150 with a focus on veterans from the Korean War. Towards the end of recruitment the protocol was revised to remove the focus on veterans from just the Korean War.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Metabolite Profiling | Up to 24 months
  Based on a single blood draw, identify metabolite biomarkers for achieving a stable target anticoagulant response among patients at a maintenance dose of warfarin.

CONTACTS AND LOCATIONS:
Overall Officials: Grover P Miller, PhD, Principal Investigator — University of Arkansas; Eugene Smith, III, MD, Principal Investigator — Dentral Arkansas Veterans Healthcare System
Locations (2):
- United States (2):
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas